CLINICAL TRIAL: NCT03511781
Title: Hypofractionated Radiotherapy Schedule of 35 Gray in 10 Fractions in Advanced Incurable Breast Cancer: A Prospective Phase I/II Study
Brief Title: Palliative Hypofractionated Radiotherapy in Advanced Incurable Breast Cancer
Acronym: HYPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC/TMC/31/14
Record Dates: First submitted 2016-10-18; First posted 2018-04-30 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Carcinoma Breast Stage IV
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm study (Experimental): Hypofractionated Radiotherapy Schedule of 35 GY in 10 fractions is being administered in advanced Incurable Breast Cancer for female patients
  Interventions: Radiation: Hypofractionated Radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated Radiotherapy — Palliative Hypofractionated radiotherapy 35 GY in 10 fractions over 2 weeks in advanced incurable Breast Cancer

SUMMARY:
This prospective phase I/II study to assess the clinical toxicity and investigate the clinical response of breast cancers to a 10 fraction hypofractionated course of radiation therapy in advanced incurable breast cancer patients. This study would also investigate the feasibility of voluntary breath hold technique for heart sparing in left sided breast cancer patients. An intervention radiation therapy dose of 35 Gray in 10 fractions over 2 weeks, 5 fractions per week, 1 fraction per day will be studied within this clinical trial. Primary objective of the study is to assess the toxicity using CTCAE version 4 and LENTSOMA toxicity criteria, in advanced incurable breast cancer patients treated with hypofractionated radiotherapy schedule of 35 GY in 10 fractions . Secondary objectives are 1. response rate after radiotherapy measured using the PERCIST criteria at 3 months. 2. Change in quality of life measured using trial outcome index (TOI) at 2 weeks after radiotherapy. 3. Measure the change in PHQ4 score at 2 weeks after radiotherapy.

Additionally to assess the feasibility of voluntary breath hold technique for heart sparing in left sided breast cancer patients and to biobank tissue and blood for future radiobiology tests. A total of 30 patients will be recruited in this study. Among these 30 patients at least 10 patients will be recruited with left sided breast cancer on which feasibility of voluntary breath hold technique for heart sparing will be tested. Patient will be followed up weekly during radiotherapy, then monthly for 1st three months, then 3 monthly for two years, then 6 monthly for next 3 years.

DETAILED DESCRIPTION:
Study design: Prospective interventional phase I/II study Study area: Tata Medical Center, Kolkata

Aims and objectives:

Primary objective To assess the toxicity using CTCAE version 4 and LENTSOMA toxicity criteria, in advanced incurable breast cancer patients treated with hypofractionated radiotherapy schedule of 35 GY in 10 fractions Secondary objectives

1. response rate after radiotherapy measured using the PERCIST criteria at 3 months. 2. Change in quality of life measured using trial outcome index (TOI) at 2 weeks after radiotherapy. 3. Measure the change in PHQ4 score at 2 weeks after radiotherapy.

To assess the impact of hypofractionated breast radiotherapy schedule of 35 GY in 10 fractions over 2 weeks on quality of life in advanced incurable breast cancer patients using FACT B scores PHQ4 questionnaire

To assess the feasibility of voluntary breath hold technique for heart sparing in left sided breast cancer patients.

To biobank tissue and blood for future radiobiology tests

Consent:

All patients will be recruited after obtaining informed consent.

Sample size:

A total of 30 patients will be recruited in this phase I/ II study. Among these 30 patients at least 10 patients will be recruited with left sided breast cancer on which feasibility of voluntary breath hold technique for heart sparing will be tested.

Statistical analysis:

Given that this is a phase I/II study a 30 patients sample is used as a feasibility study. Primary end point of this study is acute toxicity and secondary endpoint is radiological response, quality of life after radiotherapy ( from baseline) . Acute toxicities are defined as toxicities happening during and at 3 months after radiotherapy. Medcalc version 12 will be used for statistical analysis. Paired Student t test (2-tailed) was applied to compare the results from the different time points. The level of significance will be taken as P < 0.05.

Stopping Rules:

6 patients will be recruited in the first phase of the study (20% of total number). If 1-2 of the 6 patients have had more than grade 3 acute toxicity (radiation dermatitis) then the study will recruit 4 further patients as phase 2. If more than 1 of these patients are found to have more than Grade 3 dermatological toxicity then the study will be stopped. Similarly after recruitment of 20 patients, another safety monitoring will be undertaken . At any point, if more than 40% of the patients have more than grade 3 toxicity the study will be closed.

Objective Imaging in the trial:

A regional positron emission computed -computed Tomography scan of breast done before starting radiotherapy. The standardized uptake value by the tumour, size of the tumour along with that of the regional lymph nodes will be recorded. 3 months post completion of radiation, the PET-CT scan will be repeated and parameters re-recorded. PERCIST criteria will be used to evaluate response to radiation therapy.

Radiation Therapy Technique:

Acquisition of planning CT scan-

The patient is positioned supine on all in one solution breast board with head rest, arms above head as in treatment position such that the sternum is horizontal . The CT markers are placed on the patient approximately at the lower end of sternum in free breathing.The position of palpable breast tissue, drain sites and scars are marked with radio opaque wires during the CT . Helical CT scan is obtained with 5 mm thickness. Couch height from the lateral lasers are measured as reference height for reproducing in treatment table. CT marker positions are tattooed.

Acquisition of Outlines- A full 3D set of outlines covering the whole breast and the organs at risk must be collected with a slice separation of no more than 5 mm. The right breast patients are scanned with standard institutional protocol and left breast will be scanned with Voluntary breath Hold Technique . The position of palpable breast tissue, and scars are marked with radio opaque wires during the CT scan. Bolus will be used as and when required for dose build up to the surface during simulation and treatment.

Target Volume Definition-

Gross Tumour Volume (GTV)- GTV will be outlined as seen on the planning CT scan, with information available from the PET-CT scan and clinical examination. This will include any lymph nodes in the axilla or supraclavicular fossa.

Whole Breast Clinical Target Volume (WBCTV)- This is based on the recommendations in the START trial protocol . The CTV includes the soft tissues of the whole breast from 5 mm below the skin surface down to the deep fascia, excluding muscle and underlying rib cage. If the tumor is seen to involve the muscle, skin or adjoining structures adequate margins must be taken to include these in the target volume.

Planning Target Volumes (PTV)- A field-based whole breast PTV will be used and this method is illustrated below.

Intended field limits:

Breast:

1. Lateral or central tumour - Superior edge - 1cm above the superior border of the palpable breast tissue Inferior limit - 1cm below palpable breast tissue Lateral limit -1cm lateral to palpable breast, at or anterior to mid axillary line.

   Medial limit -1cm medial to palpable breast tissue at or ipsilateral to midline.

   Anterior- Adequate margin on skin anteriorly to account for respiratory movements as well as random and systematic errors
2. Medial tumour As above but medial edge may be beyond midline. The internal mammary nodes are not routinely included in the treated volume.

Supraclavicular fossa Superior: At level of cricoid or 3 cm above medial end clavicle (whichever is superior).

Inferior: Matchplane. In some patients with a lower match plane (for anatomy or mobility) Lateral: Junction of medial 2/3rd and lateral 1/3rd of the clavicle, including coracoid process

Medial: Medial margin of head of clavicle Axilla:Axilla will be included in tangential field if there is involved node clinically or radiologically in axilla.

Organs at Risk (OAR):

It is mandatory to contour ipsilateral and contralateral lung and heart, brachial plexus for dose volume histogram assessment. Left anterior descending coronary artery will be contoured for left sided breast cancer patients.

Radiotherapy planning Prescribed Dose 35 Gy in 10 fraction; 5 fractions a week; 1 fraction a day for 2 weeks. Ideally, prescribed to 100% (normalization point). Dose Planning two standard isocentric tangential fields, one lateral tangential and another medial tangential field (6 Mega Volt, 15 MV or both could be used depending on the site and geometry of the breasts) will be used to treat the breast encompassing the axillary nodes in clinically or radio-logically involved. Supraclavicular fossa will be treated with one direct anterior field. Radiotherapy will be delivered to the whole breast using tangential photons . 3D dose calculation will be done by Analytical Anisotropic Algorithm algorithm. Segmented fields with multi leaf or wedges will be used to achieve dose homogeneity in accordance with the guidelines of ICRU 50/62 i.e, within 95% to 107%. Dose reporting Tangential fields prescribed at the normalization point (ICRU reference point). The Supraclavicular field is prescribed at a depth of Dmax for 6MV beam.

Radiotherapy Treatment Setup:

Patient will be positioned in the treatment couch as in planning CT with the help of skin reference markers. The patient is then moved to planned isocenter according to the plan.The medial and lateral borders are marked and verified by light field and source-to-surface distance. The superior border of tangential fields and inferior border of supraclavicular field is matched on the skin with light field.

Radiotherapy Treatment Delivery:

After checking the alignment , the treatment commences. Every day the patient is moved from reference CT-Isocenter to planned isocenter and field edge (as defined by light field) is marked with marker at every fraction.

Planning Documentation:

Electronic Treatment prescription. Planning approval and treatment approval is given on treatment planning system. A hard copy of the planning with electronic approvals is attached with each patient file.

treatment planning system

Quality assurance and Treatment setup verification:

In-vivo dosimetry with thermoluminescence dosimeters (TLDs) and Gafchromic film will be performed during patient treatment. TLDs will be used to verify the skin dose in the junction of SCF and tangential fields and along the skin surface of intact breast for each patient for first 3 days. Film dosimetry will be used in the junction of the of Supra clavicular fossa and Tangential field. Online clinical breast coverage verification is carried out by Visually checking the light field on the patient on the first day of treatment. Partial conebeam CT scan will be taken to ascertain the treatment position verification for whole breast set-up and 2D MV image for supraclavicular field setup, for all fractions. Treatment Review Patients are reviewed weekly, unless specified otherwise by the clinician.

Dose Constraints for Organs at Risk (OAR):

The optimal dose constraints criterias are as follows-

* The volume of ipsilateral lung receiving 10.5 Gy should be less than 15%
* The volume of heart receiving 1.75 Gy and 8.75 Gy should be less than 30% and 5% respectively.
* Brachial plexus: EQD2 = 60 Gy (conservative estimate based on α/β= 2 for brachial plexus). Minimum , maximum and median dose to the left anterior descending artery will be recorded for left sided breast cancer patients undergoing voluntary breadth hold technique. In case where optimal dose constraints criteria for heart and lung could not be met in order to cover the gross tumour volume in breast or axilla; essential criteria should be met ( V10.5 Gy for lung <31%, V8.75 Gy for heart <11%).

Assessment of toxicity:

Acute toxicity will be assessed weekly during radiotherapy then monthy for 1st three month after completion of radiotherapy. Acute toxicity will be graded according to CTCAE version 4 toxicity criteria. If CTCAE Gr 3 desquamation is seen the patient will be reviewed weekly until the desquamation is resolved to CTCAE gr 1 or less. If the patient somehow fails to attend for the toxicity assessment, a telephone questionnaire will be asked to assess grade of skin toxicity. Modified LENT-SOMA scale will be used for scoring various grades of late effects occurring in brachial plexus after radiation therapy at 3 months,6 months and 1year .

Assessment of response:

Clinical assessment:

Tumour size measurement will be done pretreatment and 3 months after completion of radiotherapy. Patients will be assessed for symptoms like breast pain, ulcer, arm oedema , shoulder stiffness and others at baseline . If the patients have any of these symptoms then : for Pain in breast visual analogue scale will be used to score the pain (score 0-10), ulcer and arm oedema will be graded according to CTCAE version 4, shoulder stiffness will be recored as yes/no response. Symptom assessment will be repeated at 2 wks, 1 month, 2 months, 3 months, 6 months, and 1 year.

Radiological assessment:

All patients will have a baseline regional PET-CT scan of breast (including axilla and supraclavicular fossa) done before start of radiotherapy and three month after completion of radiotherapy another regional PET-CT scan of breast will be done. Response will be assessed using PERCIST 1.0 criteria .

Assessment of quality of life: Quality of life will be assessed by using FACT B scale and anxiety/mood symptoms will be assessed by a 4 question screen (PHQ4) before start of radiotherapy, after completion of radiotherapy and 3 month, 6 months and 1 year after completion of radiotherapy. For patients who are unable to travel, the quality of life rating will be done over telephone for the 3 months, 6 months and 1 year follow up.

Follow up:Weekly during radiotherapy, then monthly for 1st three months, then 3 monthly for two years, then 6 monthly for next 3 years.

Data Safety Monitoring An independent data safety monitoring committee (IDMC) will be instigated to monitor the progress of the trial. Two radiation oncologists, a surgeon and a lay person will be in the committee to ensure safety of patients. The IDMC will meet in confidence after a first phase of recruitment of 6 patients (20% of the sample size). The second meeting will be done after 10 patients are recruited and the third meeting after 20 patients recruited. A report of the findings and recommendations will be produced following each meeting and a summary of the minutes will be submitted to the PI, and if required, the Institutional review board.

Liability/Indemnity/Insurance:

Indemnity arrangements will be made as required.

ELIGIBILITY:
Inclusion Criteria: (all of 1-4)

1.Invasive carcinoma of the breast 2.ECOG performance Status:0,I,II 3a.Locally Advanced breast cancer which is not amenable to curative surgery as decided by Multidisciplinary tumor board OR 3b.Metastatic breast cancer patients: i) who are awaiting palliative locoregional radiotherapy for symptom (pain,bleeding,ulceration) ii) who have completed a scheduled course of palliative chemotherapy and is felt to benefit from local radiation therapy 4.Able to give consent

Exclusion Criteria:

1. Breast reconstruction using implants
2. Concurrent cyto-toxic chemotherapy -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-09; Primary Completion 2020-10 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with CTCAE 4.03 defined Grade 3 or more toxicity | 2 Years
  The proportion of patients with CTCAE 4.03 defined Grade 3 or more toxicity related to radiotherapy will be assesed. This will include toxicities like radiation fibrosis, lymphedema, pneumonitis and brachial plexopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjoy Chatterjee, FRCP,FRCR, Principal Investigator — Tata Medical Center,Kolkata
Locations (1):
- Tata Medical Center, Kolkata, West Bengal, India

IPD SHARING:
Plan to Share IPD: Undecided
Once appropriate authorities approach and once clearance of local authorities is received, data could be shared

REFERENCES:
- [Background] Clarke M, Collins R, Darby S, Davies C, Elphinstone P, Evans V, Godwin J, Gray R, Hicks C, James S, MacKinnon E, McGale P, McHugh T, Peto R, Taylor C, Wang Y; Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of radiotherapy and of differences in the extent of surgery for early breast cancer on local recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 Dec 17;366(9503):2087-106. doi: 10.1016/S0140-6736(05)67887-7. PMID 16360786
- [Background] Darby SC, Ewertz M, McGale P, Bennet AM, Blom-Goldman U, Bronnum D, Correa C, Cutter D, Gagliardi G, Gigante B, Jensen MB, Nisbet A, Peto R, Rahimi K, Taylor C, Hall P. Risk of ischemic heart disease in women after radiotherapy for breast cancer. N Engl J Med. 2013 Mar 14;368(11):987-98. doi: 10.1056/NEJMoa1209825. PMID 23484825